CLINICAL TRIAL: NCT02346240
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo- and Active-Controlled Study Followed by a Placebo-Controlled Maintenance Period and Open-Label Follow-Up to Evaluate the Efficacy and Safety of Certolizumab Pegol in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety Study of Certolizumab Pegol (CZP) Versus Active Comparator and Placebo in Subjects With Plaque Psoriasis (PSO)
Acronym: CIMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0003; 2014-003492-36 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: Certolizumab Pegol; Cimzia; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Certolizumab Pegol; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CZP 200 mg (Experimental): Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg at Weeks 0, 2, 4, followed by CZP 200 mg every two weeks (Q2W) from Week 6 to Week 14.
  The treatment received from Week 16 to Week 48 is based on initial treatment and response to treatment at Week 16:
  * Subjects with a PASI75 response at Week 16 will be re-randomized to receive either CZP 200 mg Q2W or CZP 400 mg every 4 weeks (Q4W; with Placebo administered on alternate dosing weeks to maintain the blind) or Placebo Q2W.
  * Subjects who do not achieve a PASI75 response at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  Subjects can enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Interventions: Biological: Certolizumab Pegol
- CZP 400 mg (Experimental): Certolizumab Pegol subcutaneous (sc) injection 400 mg every two weeks (Q2W) through Week 14.
  The treatment received from Week 16 to Week 48 is based on initial treatment and response to treatment at Week 16:
  * Subjects with a PASI75 response at Week 16 will be re-randomized to CZP 200 mg Q2W or CZP 400 mg Q2W or Placebo Q2W.
  * Subjects who do not achieve a PASI75 response at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  Subjects can enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Interventions: Biological: Certolizumab Pegol
- Etanercept (Active Comparator): Etanercept (ETN) subcutaneous (sc) injection 50 mg twice weekly through Week 12.
  The treatment received from Week 16 to Week 48 is based on initial treatment and response to treatment at Week 16:
  * Subjects with a PASI75 response at Week 16 will be re-randomized to either Certolizumab Pegol (loading dose of 400 mg at Weeks 16, 18, and 20 followed by 200 mg Q2W) or Placebo Q2W.
  * Subjects who do not achieve a PASI75 response at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  Subjects can enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Interventions: Biological: Etanercept
- Placebo (Placebo Comparator): Placebo subcutaneous (sc) injection every two weeks (Q2W).
  The treatment received from Week 16 to Week 48 is based on initial treatment and response to treatment at Week 16:
  * Subjects with a PASI75 response at Week 16 continue to receive blinded Placebo.
  * Subjects who do not achieve a PASI75 response at Week 16 will be removed from blinded study medication and escape to CZP 400 mg Q2W. Subjects who receive unblinded CZP 400 mg Q2W for 16 weeks and do not achieve a PASI50 response will be withdrawn from the study.
  Subjects can enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 200 mg/ mL
  * Route of Administration: Subcutaneous use
  Other Names: Cimzia; CDP870; CZP
  Arms: CZP 200 mg; CZP 400 mg
Biological: Etanercept — * Active Substance: Etanercept
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 50 mg / mL
  * Route of Administration: Subcutaneous use
  Other Names: Enbrel; ETN
  Arms: Etanercept
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 0.9 % saline
  * Route of Administration: Subcutaneous use
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of two dose levels of certolizumab pegol compared to active comparator and placebo in adults with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
This study consists of the following Periods:

* Initial Treatment Period from Week 0 to Week 16
* Maintenance Treatment Period from Week 16 to Week 48
* Open-label Extension Treatment Period (96 weeks)
* Safety Follow-Up (10 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Adult men or women >= 18 years
* Chronic plaque psoriasis for at least 6 months
* Baseline psoriasis activity and severity index >= 12 and body surface area >= 10 % and Physician's Global Assessments score >= 3
* Candidate for systemic psoriasis therapy and/or phototherapy and/or chemophototherapy
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Erythrodermic, guttate, generalized pustular form of psoriasis
* History of current, chronic, or recurrent infections of viral, bacterial, or fungal origin as described in the protocol
* Congestive heart failure
* History of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease
* Concurrent malignancy or a history of malignancy as described in the protocol
* History of, or suspected, demyelinating disease of the central nervous system (e.g., multiple sclerosis or optic neuritis)
* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 5 months following last dose of study drug in the UK, Czech Republic, Germany, and France, and within 3 months for all other countries. Male subjects who are planning a partner pregnancy during the study or within 5 months following the last dose in France and within 10 weeks in all other countries
* Any other condition which, in the Investigator's judgment, would make the subject unsuitable for participation in the study
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2015-02-11; Primary Completion 2016-03-22 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (70):
- United States (19):
  - Ps0003 317, Mobile, Alabama
  - Ps0003 306, Little Rock, Arkansas
  - Ps0003 301, Beverly Hills, California
  - Ps0003 307, Los Angeles, California
  - Ps0003 405, San Diego, California
  - Ps0003 316, Washington D.C., District of Columbia
  - Ps0003 304, West Palm Beach, Florida
  - Ps0003 302, Springfield, Illinois
  - Ps0003 313, West Dundee, Illinois
  - Ps0003 310, Indianapolis, Indiana
  - Ps0003 400, Henderson, Nevada
  - Ps0003 319, Verona, New Jersey
  - Ps0003 404, Buffalo, New York
  - Ps0003 407, Portland, Oregon
  - Ps0003 309, Johnston, Rhode Island
  - Ps0003 401, Dallas, Texas
  - Ps0003 403, Houston, Texas
  - Ps0003 406, San Antonio, Texas
  - Ps0003 311, Webster, Texas
- Bulgaria (4):
  - Ps0003 345, Dupnitsa, Kyustendil
  - Ps0003 343, Sofia, Sofia-Grad
  - Ps0003 344, Plovdiv
  - Ps0003 342, Varna
- Czechia (4):
  - Ps0003 353, Pardubice, District of Columbia
  - Ps0003 351, Pardubice
  - Ps0003 352, Prague
  - Ps0003 350, Ústí nad Labem
- France (2):
  - Ps0003 320, Nice
  - Ps0003 325, Toulouse
- Germany (15):
  - Ps0003 374, Friedrichshafen, Baden-Wurttemberg
  - Ps0003 373, Munich, Bavaria
  - Ps0003 368, Frankfurt am Main, Hesse
  - Ps0003 378, Bochum, North Rhine-Westphalia
  - Ps0003 371, Wuppertal, North Rhine-Westphalia
  - Ps0003 370, Mainz, Rhineland-Palatinate
  - Ps0003 365, Kiel, Schleswig-Holstein
  - Ps0003 363, Erfurt, Thuringia
  - Ps0003 367, Berlin
  - Ps0003 372, Berlin
  - Ps0003 375, Berlin
  - Ps0003 369, Dresden
  - Ps0003 361, Giessen
  - Ps0003 362, Hamburg
  - Ps0003 366, Hanover
- Hungary (5):
  - Ps0003 381, Orosháza, Bekes County
  - Ps0003 380, Debrecen, Hajdú-Bihar
  - Ps0003 382, Budapest
  - Ps0003 383, Budapest
  - Ps0003 384, Budapest
- Ps0003 340, Breda, Netherlands
- Poland (14):
  - Ps0003 424, Poznan, Greater Poland Voivodeship
  - Ps0003 330, Torun, Kuyavian-Pomeranian Voivodeship
  - Ps0003 422, Wroclaw, Lower Silesian Voivodeship
  - Ps0003 335, Lublin, Lublin Voivodeship
  - Ps0003 338, Warsaw, Masovian Voivodeship
  - Ps0003 421, Warsaw, Masovian Voivodeship
  - Ps0003 333, Bialystok, Podlaskie Voivodeship
  - Ps0003 334, Katowice, Silesian Voivodeship
  - Ps0003 425, Bialystok
  - Ps0003 427, Gdansk
  - Ps0003 423, Gdynia
  - Ps0003 332, Szczecin
  - Ps0003 336, Warsaw
  - Ps0003 339, Wroclaw
- United Kingdom (6):
  - Ps0003 390, Dundee, Angus
  - Ps0003 391, Hexham, Northumberland
  - Ps0003 395, Cardiff, Wales
  - Ps0003 393, Edgbaston
  - Ps0003 394, Liverpool
  - Ps0003 392, Manchester

REFERENCES:
- [Result] Lebwohl M, Blauvelt A, Paul C, Sofen H, Weglowska J, Piguet V, Burge D, Rolleri R, Drew J, Peterson L, Augustin M. Certolizumab pegol for the treatment of chronic plaque psoriasis: Results through 48 weeks of a phase 3, multicenter, randomized, double-blind, etanercept- and placebo-controlled study (CIMPACT). J Am Acad Dermatol. 2018 Aug;79(2):266-276.e5. doi: 10.1016/j.jaad.2018.04.013. Epub 2018 Apr 14. PMID 29660425
- [Result] Warren RB, Lebwohl M, Sofen H, Piguet V, Augustin M, Brock F, C Arendt, Fierens F, Blauvelt A. Three-year efficacy and safety of certolizumab pegol for the treatment of plaque psoriasis: results from the randomized phase 3 CIMPACT trial. J Eur Acad Dermatol Venereol. 2021 Dec;35(12):2398-2408. doi: 10.1111/jdv.17486. Epub 2021 Aug 17. PMID 34192387
- [Derived] Blauvelt A, Paul C, van de Kerkhof P, Warren RB, Gottlieb AB, Langley RG, Brock F, Arendt C, Boehnlein M, Lebwohl M, Reich K. Long-term safety of certolizumab pegol in plaque psoriasis: pooled analysis over 3 years from three phase III, randomized, placebo-controlled studies. Br J Dermatol. 2021 Apr;184(4):640-651. doi: 10.1111/bjd.19314. Epub 2020 Sep 6. PMID 32531798
- See also: Related Info — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll participants in February 2015, from multiple sites in Europe and United States and concluded in December 2018. 559 participants are included in the Randomized Set (RS) shown in the Participant Flow.
Pre-assignment Details: The study included a Screening Period, an Initial Treatment Period up to Week 16, a Maintenance Treatment Period up to Week 48, an Open-Label Extension Treatment Period up to Week 144 and a Safety Follow-up Period up to Week 157. The Participants Flow refers to the Randomized Set, the Maintenance Set and the Open Label Set.
Groups:
- Placebo Q2W: Placebo subcutaneous (sc) injections every 2 weeks (Q2W) through Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 continued to receive blinded Placebo. PASI75 non-responders at Week 16 were removed from blinded study medication and escaped to Certolizumab pegol (CZP) 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  Participants could enter a 96-week open-label extension period after completing the Maintenance Period (Weeks 16-48) and receive CZP under certain conditions.
- Etanercept: Etanercept (ETN) 50 mg subcutaneous (sc) injections twice per week throughout Week 11.5.
  •PASI75 responders at Week 16 were re-randomized to either CZP (loading dose of 400 mg at Weeks 16, 18, and 20 followed by 200 mg Q2W) or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
- CZP 200 mg Q2W: CZP 400 mg injections at Weeks 0, 2, 4, followed by CZP 200 mg every 2 weeks (Q2W) from Week 6 to Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 were re-randomized to receive either CZP 200 mg Q2W or CZP 400 mg every 4 weeks (Q4W); with Placebo administered on alternate dosing weeks to maintain the blind) Or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 were removed from blinded study medication and escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
- CZP 400 mg Q2W: CZP 400 mg injections every 2 weeks (Q2W) through Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 were re-randomized to CZP 200 mg Q2W or CZP 400 mg Q2W or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 were removed from blinded study medication and escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
- Placebo/Placebo Q2W: This arm consisted of participants initially randomized in the Placebo arm, who achieved a PASI75 response at Week 16 and continued to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48).
- Etanercept/Placebo Q2W: This arm consisted of participants initially randomized in the Etanercept arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48).
- Etanercept/CZP 200 mg Q2W: This arm consisted of participants initially randomized in the Etanercept arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48).
- CZP 200 mg Q2W/Placebo Q2W: This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48).
- CZP 200 mg Q2W/CZP 200 mg Q2W: This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48).
- CZP 200 mg Q2W/CZP 400 mg Q4W: This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 400 mg Q4W in the Maintenance Period (Week 16 to Week 48).
- CZP 400 mg Q2W/Placebo Q2W: This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48).
- CZP 400 mg Q2W/CZP 200 mg Q2W: This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48).
- CZP 400 mg Q2W/CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 400 mg Q2W in the Maintenance Period (Week 16 to Week 48).
- Placebo Q2W/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the Placebo arm, who did not achieve a PASI75 response at Week 16 escaped from the blinded treatment and received CZP 400 mg every two weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- Etanercept/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the Etanercept arm, who did not achieve a PASI75 response at Week 16 escaped from the treatment and received CZP 400 mg every two weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- CZP 200 mg Q2W/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 200 mg arm, who did not achieve a PASI75 response at Week 16 escaped from the blinded treatment and received CZP 400 mg every two weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- CZP 400 mg Q2W/Escape CZP 400 mg Q2W: This arm consisted of participants initially randomized in the CZP 400 mg arm, who did not achieve a PASI75 response at Week 16 escaped from the blinded treatment and received CZP 400 mg every two weeks. Participants who did not achieve PASI50 after 16 weeks of unblinded treatment were withdrawn from the study.
- Placebo/CZP 200 mg Q2W OLE: This arm consisted of participants from the Placebo-controlled Maintenance Period, who achieved PASI50 response (had no relapse) at Week 48 and entered the 96-Weeks OLE Period receiving CZP 200 mg Q2W.
- CZP 200 mg Q2W/CZP 200 mg Q2W OLE: This arm consisted of participants who received CZP 200 mg Q2W in the Maintenance Period, who achieved a PASI50 response (had no relapse) at Week 48 and entered OLE.
- CZP 400 mg Q4W/CZP 200 mg Q2W OLE: This arm consisted of participants who received CZP 400 mg Q4W in the Maintenance Period, who achieved a PASI50 response (had no relapse) at Week 48 and entered OLE on the CZP 200mg Q2W dose.
- CZP 400 mg Q2W/CZP 200 mg Q2W OLE: This arm consisted of participants who received CZP 400 mg Q2W in the Maintenance Period, who achieved a PASI50 response (had no relapse) at Week 48 and entered OLE on the CZP 200mg Q2W dose.
- Esc CZP 400 mg Q2W/CZP 400 mg Q2W OLE: This arm consisted of participants who received open-label CZP 400mg Q2W in the Maintenance Period and entered OLE.
- Placebo/CZP 400 mg Q2W OLE: This arm consisted of participants from the Placebo-controlled Maintenance Period, who did not achieve PASI50 response (had relapse) and entered the 96-weeks OLE Period receiving CZP 400 mg Q2W.
- Any CZP/CZP 400 mg Q2W OLE: This arm consisted of participants who relapsed on CZP 200 mg Q2W, CZP 400 mg Q4W and 400 mg Q2W.
Period: Initial Period (Baseline to Week 16)
Arm/Group | Placebo Q2W | Etanercept | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Etanercept/Placebo Q2W | Etanercept/CZP 200 mg Q2W | CZP 200 mg Q2W/Placebo Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 400 mg Q4W | CZP 400 mg Q2W/Placebo Q2W | CZP 400 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo Q2W/Escape CZP 400 mg Q2W | Etanercept/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q4W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Esc CZP 400 mg Q2W/CZP 400 mg Q2W OLE | Placebo/CZP 400 mg Q2W OLE | Any CZP/CZP 400 mg Q2W OLE
Started | 57 | 170 | 165 | 167 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 55 | 159 | 159 | 162 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Finished Wk16 Started Maintenance Period | 55 | 159 | 159 | 160 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 55 | 159 | 159 | 160 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 11 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject missed 3 visits | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16 to Week 48)
Arm/Group | Placebo Q2W | Etanercept | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Etanercept/Placebo Q2W | Etanercept/CZP 200 mg Q2W | CZP 200 mg Q2W/Placebo Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 400 mg Q4W | CZP 400 mg Q2W/Placebo Q2W | CZP 400 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo Q2W/Escape CZP 400 mg Q2W | Etanercept/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q4W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Esc CZP 400 mg Q2W/CZP 400 mg Q2W OLE | Placebo/CZP 400 mg Q2W OLE | Any CZP/CZP 400 mg Q2W OLE
Started | 0 | 0 | 0 | 0 | 2 | 24 | 50 | 22 | 44 | 44 | 25 | 50 | 49 | 53 | 85 | 49 | 36 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Maintenance Period | 0 | 0 | 0 | 0 | 2 | 23 | 48 | 20 | 40 | 43 | 23 | 47 | 49 | 46 | 71 | 36 | 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Finished Wk48 Entered Open-label Period | 0 | 0 | 0 | 0 | 2 | 23 | 48 | 20 | 40 | 43 | 23 | 47 | 49 | 45 | 68 | 35 | 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 23 | 48 | 20 | 40 | 43 | 23 | 47 | 49 | 45 (1 subject completed the Maintenance Period but did not enter the Open-Label Period.) | 68 (3 subjects completed the Maintenance Period but did not enter the Open-Label Period.) | 35 (1 subject completed the Maintenance Period but did not enter the Open-Label Period.) | 29 (1 subject completed the Maintenance Period but did not enter the Open-Label Period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 1 | 2 | 3 | 0 | 8 | 17 | 14 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not achieve PASI50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Moved out of state | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision due to non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse events and alcohol problem | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient's decisions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unavailability due to business trip | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient request due to non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period (Week 48 to Week 144)
Arm/Group | Placebo Q2W | Etanercept | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo Q2W | Etanercept/Placebo Q2W | Etanercept/CZP 200 mg Q2W | CZP 200 mg Q2W/Placebo Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 400 mg Q4W | CZP 400 mg Q2W/Placebo Q2W | CZP 400 mg Q2W/CZP 200 mg Q2W | CZP 400 mg Q2W/CZP 400 mg Q2W | Placebo Q2W/Escape CZP 400 mg Q2W | Etanercept/Escape CZP 400 mg Q2W | CZP 200 mg Q2W/Escape CZP 400 mg Q2W | CZP 400 mg Q2W/Escape CZP 400 mg Q2W | Placebo/CZP 200 mg Q2W OLE | CZP 200 mg Q2W/CZP 200 mg Q2W OLE | CZP 400 mg Q4W/CZP 200 mg Q2W OLE | CZP 400 mg Q2W/CZP 200 mg Q2W OLE | Esc CZP 400 mg Q2W/CZP 400 mg Q2W OLE | Placebo/CZP 400 mg Q2W OLE | Any CZP/CZP 400 mg Q2W OLE
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 122 | 41 | 48 | 177 | 34 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 105 | 34 | 45 | 146 | 27 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 17 | 7 | 3 | 31 | 7 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 3 | 13 | 3 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 10 | 1 | 1
Not completed — No PASI50 response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 2 | 3
Not completed — No efficacy of study medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set consisting of all participants randomized into the study.
Arm/Group | Placebo Q2W | Etanercept | CZP 200 mg Q2W | CZP 400 mg Q2W | Total Title
Number analyzed (Participants) | 57 | 170 | 165 | 167 | 559
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 2 | 3
  Between 18 and 65 years | 53 | 156 | 153 | 154 | 516
  >=65 years | 4 | 13 | 12 | 11 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.5) | 44.6 (14.1) | 46.7 (13.5) | 45.4 (12.4) | 45.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 43 | 52 | 60 | 178
  Male | 34 | 127 | 113 | 107 | 381
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 3 | 3 | 7
  Black or African American | 0 | 3 | 2 | 2 | 7
  White | 57 | 163 | 158 | 162 | 540
  Other/mixed | 0 | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI75) Response at Week 12
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: The Randomized Set (RS) consisted of all participants randomized into the study.
  Missing data were handled using the Markov Chain Monte Carlo (MCMC) method for multiple imputation.
Measure: Number; unit: percentage of participants
Groups:
- Placebo Q2W (RS): Placebo subcutaneous (sc) injections every 2 weeks (Q2W) through Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 continued to receive blinded Placebo. PASI75 non-responders at Week 16 were removed from blinded study medication and escaped to Certolizumab pegol (CZP) 400 mg Q2W. Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study.
  Participants could enter a 96-week open-label extension period after completing the Maintenance Period (Weeks 16-48) and receive CZP under certain conditions.
  Participants formed the Randomized Set (RS).
- Etanercept (RS): Etanercept (ETN) 50 mg subcutaneous (sc) injections twice per week throughout Week 11.5.
  •PASI75 responders at Week 16 were re-randomized to either CZP (loading dose of 400 mg at Weeks 16, 18, and 20 followed by 200 mg Q2W) or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Participants formed the Randomized Set (RS).
- CZP 200 mg Q2W (RS): CZP 400 mg injections at Weeks 0, 2, 4, followed by CZP 200 mg every 2 weeks (Q2W) from Week 6 to Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 were re-randomized to receive either CZP 200 mg Q2W or CZP 400 mg every 4 weeks (Q4W); with Placebo administered on alternate dosing weeks to maintain the blind) Or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 were removed from blinded study medication and escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Participants formed the Randomized Set (RS).
- CZP 400 mg Q2W (RS): CZP 400 mg injections every 2 weeks (Q2W) through Week 14. Treatment received from Week 16-48 is based on initial treatment and response to treatment:
  •PASI75 responders at Week 16 were re-randomized to CZP 200 mg Q2W or CZP 400 mg Q2W or Placebo Q2W. Participants who did not achieve a PASI75 response at Week 16 were removed from blinded study medication and escaped to CZP 400 mg Q2W.
  Participants who received unblinded CZP 400 mg Q2W for 16 weeks and did not achieve a PASI50 response were withdrawn from the study. Participants could enter a 96-week open-label extension period after completing the Maintenance Period and receive CZP under certain conditions.
  Participants formed the Randomized Set (RS).
Arm/Group | Placebo Q2W (RS) | Etanercept (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 170 | 165 | 167
percentage of participants | 5.0 | 53.3 | 61.3 | 66.7
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); The statistical analysis of the co-primary efficacy variables and key secondary efficacy variables accounted for multiplicity by using a fixed sequence testing procedure; Test type: Superiority; Regression, Logistic; Estimated responder rate, CIs, p-values based on a logistic regression model with factors for treatment, region, prior biologic exposure; Estimated difference in responder rate = 61.6, 95% CI 2-sided [52.1 to 71.2] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 56.2, 95% CI 2-sided [46.4 to 66.0] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; Odds ratios, CIs, p-values based on a logistic regression model with factors for treatment, region, prior biologic exposure; Odds Ratio (OR) = 37.988, 95% CI 2-sided [11.312 to 127.576]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 30.023, 95% CI 2-sided [8.971 to 100.481]
Statistical Analysis 5: Comparison: Etanercept (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 13.4, 95% CI 2-sided [2.7 to 24.1] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Etanercept Q2W (RS)
Statistical Analysis 6: Comparison: Etanercept (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 8.0, 95% CI 2-sided [-2.9 to 18.9] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Etanercept Q2W (RS)
Statistical Analysis 7: Comparison: Etanercept (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0152, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. ETN; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 1.756, 95% CI 2-sided [1.114 to 2.768]
Statistical Analysis 8: Comparison: Etanercept (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1523, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. ETN; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 1.388, 95% CI 2-sided [0.886 to 2.175]

2. Secondary Outcome: Proportion of Subjects Who Achieve a Physician's Global Assessment (PGA) Clear or Almost Clear Response (With at Least 2 Category Improvement) at Week 12
Description: The Investigator assessed the overall severity of Psoriasis (PSO) using the following 5-point scale: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | Etanercept (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 170 | 165 | 167
percentage of participants | 1.9 | 39.2 | 39.8 | 50.3
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 48.5, 95% CI 2-sided [39.33 to 57.63] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 37.9, 95% CI 2-sided [28.88 to 46.96] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 56.129, 95% CI 2-sided [7.787 to 404.555]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0004, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 36.566, 95% CI 2-sided [5.061 to 264.196]

3. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI90) Response at Week 12
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | Etanercept (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 170 | 165 | 167
percentage of participants | 0.2 | 27.1 | 31.2 | 34.0
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 33.8, 95% CI 2-sided [20.68 to 46.98] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 31.0, 95% CI 2-sided [18.18 to 43.80] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 39.949, 95% CI 2-sided [8.407 to 189.828]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 35.084, 95% CI 2-sided [7.363 to 167.179]

4. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI75) Response at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 165 | 167
percentage of participants | 3.8 | 68.2 | 74.7
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 70.9, 95% CI 2-sided [62.15 to 79.59] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 64.4, 95% CI 2-sided [55.12 to 73.63] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 76.277, 95% CI 2-sided [17.952 to 324.094]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 55.413, 95% CI 2-sided [13.135 to 233.782]

5. Secondary Outcome: Proportion of Subjects Who Achieve a Physician's Global Assessment (PGA) Clear or Almost Clear Response (With at Least 2 Category Improvement) at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 165 | 167
percentage of participants | 3.4 | 48.3 | 58.4
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 55.0, 95% CI 2-sided [45.59 to 64.35] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 44.9, 95% CI 2-sided [35.39 to 54.49] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 40.717, 95% CI 2-sided [9.741 to 170.198]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 27.165, 95% CI 2-sided [6.504 to 113.453]

6. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI90) Response at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W (RS) | CZP 200 mg Q2W (RS) | CZP 400 mg Q2W (RS)
Number analyzed (Participants) | 57 | 165 | 167
percentage of participants | 0.3 | 39.8 | 49.1
Statistical Analysis 1: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 48.8, 95% CI 2-sided [34.22 to 63.41] — Estimate and 95 % CI for difference in proportion of responders for CZP 400 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 2: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 39.5, 95% CI 2-sided [25.58 to 53.38] — Estimate and 95 % CI for difference in proportion of responders for CZP 200 mg Q2W (RS) versus Placebo Q2W (RS)
Statistical Analysis 3: Comparison: Placebo Q2W (RS) vs CZP 400 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 400 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 72.278, 95% CI 2-sided [14.650 to 356.602]
Statistical Analysis 4: Comparison: Placebo Q2W (RS) vs CZP 200 mg Q2W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value is evaluated at a 2-sided significance level for CZP 200 mg vs. PBO; [statistical method as in outcome 1, analysis 3]; Odds Ratio (OR) = 49.527, 95% CI 2-sided [10.002 to 245.256]

7. Secondary Outcome: Proportion of Subjects Who Achieve a Psoriasis Activity and Severity Index (PASI75) Response at Week 48 for Those Achieving PASI75 at Week 16
Description: as for outcome 1
Time Frame: Week 48
Population: The Week 16 Randomized Set (WK16RS) consisted of all participants who achieved a PASI75 response at Week 16 and were re-randomized into the double-blind, placebo-controlled Maintenance Treatment Period.
  Missing data were handled using non-response imputation (NRI) methods.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Placebo Q2W (WK16RS): This arm consisted of participants initially randomized in the Placebo arm, who achieved a PASI75 response at Week 16 and continued to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- Etanercept/Placebo Q2W (WK16RS): This arm consisted of participants initially randomized in the Etanercept arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- Etanercept/CZP 200 mg Q2W (WK16RS): This arm consisted of participants initially randomized in the Etanercept arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 200 mg Q2W/Placebo Q2W (WK16RS): This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 200 mg Q2W/CZP 200 mg Q2W (WK16RS): This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 200 mg Q2W/CZP 400 mg Q4W (WK16RS): This arm consisted of participants initially randomized in the CZP 200 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 400 mg Q4W in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 400 mg Q2W/Placebo Q2W (WK16RS): This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded Placebo in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 400 mg Q2W/CZP 200 mg Q2W (WK16RS): This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 200 mg Q2W in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
- CZP 400 mg Q2W/CZP 400 mg Q2W (WK16RS): This arm consisted of participants initially randomized in the CZP 400 mg arm, who achieved a PASI75 response at Week 16 and were re-randomized to receive blinded CZP 400 mg Q2W in the Maintenance Period (Week 16 to Week 48). Participants formed the Week 16 Randomized Set (WK16RS).
Arm/Group | Placebo/Placebo Q2W (WK16RS) | Etanercept/Placebo Q2W (WK16RS) | Etanercept/CZP 200 mg Q2W (WK16RS) | CZP 200 mg Q2W/Placebo Q2W (WK16RS) | CZP 200 mg Q2W/CZP 200 mg Q2W (WK16RS) | CZP 200 mg Q2W/CZP 400 mg Q4W (WK16RS) | CZP 400 mg Q2W/Placebo Q2W (WK16RS) | CZP 400 mg Q2W/CZP 200 mg Q2W (WK16RS) | CZP 400 mg Q2W/CZP 400 mg Q2W (WK16RS)
Number analyzed (Participants) | 2 | 24 | 50 | 22 | 44 | 44 | 25 | 50 | 49
percentage of participants | 100 | 8.3 | 82.0 | 45.5 | 79.5 | 88.6 | 36.0 | 80.0 | 98.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) until Week 144.
Description: At Week 16, only 2 participants continued PBO until Week 48 (no patient received PBO post Week 48) and all ETN-randomized participants switched to PBO (24) or CZP (135), leading to a significantly lower exposure in PBO/ETN arms than in CZP arms.
Groups:
- Placebo Q2W (SS) Wk 0-48: This arm consisted of all participants who received Placebo (PBO) at any time in the study (Week 0 to Week 48).
  Only 2 participants received PBO from Week 16 to Week 48. Participants formed the Safety Set (SS).
- Etanercept (SS) Wk 0-12: This arm consisted of all participants who received Etanercept at any time in the study (Week 0 to Week 12).
  Participants formed the SS.
- CZP 200 mg Q2W (SS) Wk 0-144: This arm consisted of all participants who received CZP 200 mg Q2W at any time in the study (Week 0 to Week 144).
  Participants formed the SS.
- CZP 400 mg Q2W (SS) Wk 0-144: This arm consisted of all participants who received CZP 400 mg Q2W at any time in the study (Week 0 to Week 144).
  Participants formed the SS.
- CZP 400mg Q4W (SS) Wk 16-48: This arm consisted of all participants who received CZP 400 mg Q4W at any time in the study (Week 16 to Week 48).
  Participants formed the SS.
Arm/Group | Placebo Q2W (SS) Wk 0-48 | Etanercept (SS) Wk 0-12 | CZP 200 mg Q2W (SS) Wk 0-144 | CZP 400 mg Q2W (SS) Wk 0-144 | CZP 400mg Q4W (SS) Wk 16-48
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/168 | 2/373 | 1/412 | 0/44
Serious Adverse Events (participants affected / at risk) | 8/128 | 1/168 | 34/373 | 51/412 | 5/44
Other Adverse Events (participants affected / at risk) | 42/128 | 37/168 | 139/373 | 158/412 | 11/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (SS) Wk 0-48 (N=128) | Etanercept (SS) Wk 0-12 (N=168) | CZP 200 mg Q2W (SS) Wk 0-144 (N=373) | CZP 400 mg Q2W (SS) Wk 0-144 (N=412) | CZP 400mg Q4W (SS) Wk 16-48 (N=44)
Intracardiac mass (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
House dust allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium tuberculosis complex test negative (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaplastic oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Primary progressive multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (SS) Wk 0-48 (N=128) | Etanercept (SS) Wk 0-12 (N=168) | CZP 200 mg Q2W (SS) Wk 0-144 (N=373) | CZP 400 mg Q2W (SS) Wk 0-144 (N=412) | CZP 400mg Q4W (SS) Wk 16-48 (N=44)
Nasopharyngitis (Infections and infestations) | 15 (16) | 14 (14) | 56 (81) | 66 (83) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 13 (15) | 12 (14) | 38 (55) | 45 (64) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 23 (34) | 11 (13) | 2 (4)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2) | 9 (10) | 12 (13) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 14 (17) | 18 (20) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 10 (10) | 20 (23) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 3 (4) | 19 (19) | 24 (24) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days